CLINICAL TRIAL: NCT03921944
Title: Evaluation of Structural and Functional Integrity of the Rotator Cuff After Total Shoulder Arthroplasty
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, April Armstrong, Professor of Surgery, Orthopaedics, Penn State Health Milton S Hershey Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00008095
Record Dates: First submitted 2019-02-27; First posted 2019-04-19 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Osteoarthritis of Shoulder
Keywords: shoulder surgery; arthritis; rotator cuff
MeSH Terms: conditions — Arthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- total shoulder replacement surgery (Other): Subjects will be assessed for the outcome measures at one year and two year timepoints post total shoulder replacement surgery
  Interventions: Diagnostic Test: CT scan of the shoulders

INTERVENTIONS:
Diagnostic Test: CT scan of the shoulders — studies of both operative and nonoperative shoulders
  Other Names: EMG of the shoulders

SUMMARY:
The purpose of this study is to examine the rotator cuff muscles in your shoulder at one and two year post total shoulder replacement surgery.

ELIGIBILITY:
Inclusion Criteria:

* age >45yrs
* primary diagnosis of osteoarthritis of the shoulder
* total shoulder replacement performed by Dr. Armstrong
* administered a local anesthetic mixture and not regional anesthesia
* all genders
* Fluent in written and spoken English
* Patients capable of giving informed consent

Exclusion Criteria:

* Known contraindications to CT/EMG
* Inability to provide informed consent
* History of recent trauma to the shoulder
* Atypical shoulder pain
* Other suspected shoulder pathology (i.e. tumor, infection)
* Pregnancy
* Bilateral total shoulder arthroplasty

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-05-02 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Active Nerve Denervation | one year post surgery
  EMG examination will be performed by a single neurologist. The EMG Examination will be performed on the muscles (upper subscapularis, supraspinatus, infraspinatus, teres minor and rhomboid) to look for any presence or absence of active denervation. Presence indicated by increased insertional activity, fibrillation potential, positive sharp waves and/or with fasciculations in both operated and unoperated shoulders.
Active Nerve Denervation | two year post surgery
  EMG examination will be performed by a single neurologist. The EMG Examination will be performed on the muscles (upper subscapularis, supraspinatus, infraspinatus, teres minor and rhomboid) to look for any presence or absence of active denervation. Presence indicated by increased insertional activity, fibrillation potential, positive sharp waves and/or with fasciculations in both operated and unoperated shoulders.
Neuropathic Changes_amplitude | one year post surgery
  The EMG Examination will be performed on the muscles (upper subscapularis, supraspinatus, infraspinatus, teres minor and rhomboid) to look for the presence or absence of neuropathic changes assessed by examining unit morphology amplitude: measured in millivolts, in both operated and unoperated shoulders.
Neuropathic Changes_amplitude | two year post surgery
  The EMG Examination will be performed on the muscles (upper subscapularis, supraspinatus, infraspinatus, teres minor and rhomboid) to look for the presence or absence of neuropathic changes assessed by examining unit morphology amplitude: measured in millivolts, in both operated and unoperated shoulders.
Neuropathic Changes_recruitment pattern | one year post surgery
  The EMG Examination will be performed on the muscles (upper subscapularis, supraspinatus, infraspinatus, teres minor and rhomboid) to look for the presence or absence of neuropathic changes assessed by examining unit morphology: phases with recruitment pattern measured as 1-2 or 3-4 units in both operated and unoperated shoulders.
Neuropathic Changes_recruitment pattern | two year post surgery
  The EMG Examination will be performed on the muscles (upper subscapularis, supraspinatus, infraspinatus, teres minor and rhomboid) to look for the presence or absence of neuropathic changes assessed by examining unit morphology: phases with recruitment pattern measured as 1-2 or 3-4 units in both operated and unoperated shoulders.
Neuropathic Changes_duration | one year post surgery
  The EMG Examination will be performed on the muscles in both operated and unoperated shoulders to look for the presence or absence of neuropathic changes assessed by examining unit morphology: duration measured in milliseconds.
Neuropathic Changes_duration | two year post surgery
  The EMG Examination will be performed on the muscles in both operated and unoperated shoulders to look for the presence or absence of neuropathic changes assessed by examining unit morphology: duration measured in milliseconds.
Total number of Muscles affected with active denervation | one year post surgery
  The EMG Examination will be performed to look for abnormal changes as indicated by presence of active nerve denervation across the 5 muscles (upper subscapularis, Infraspinatus, Supraspinatus, teres minor, Rhomboid) in both operated and unoperated shoulders.
Total number of Muscles affected with active denervation | two year post surgery
  The EMG Examination will be performed to look for abnormal changes as indicated by presence of active nerve denervation across the 5 muscles (upper subscapularis, Infraspinatus, Supraspinatus, teres minor, Rhomboid) in both operated and unoperated shoulders.
Total number of muscles affected with neuropathic changes | one year post surgery
  The EMG Examination will be performed to look for neuropathic changes as indicated by amplitude, recruitment pattern and duration across the 5 muscles (upper subscapularis, Infraspinatus, Supraspinatus, teres minor, Rhomboid) in both operated and unoperated shoulders.
Total number of muscles affected with neuropathic changes | two year post surgery
  The EMG Examination will be performed to look for neuropathic changes as indicated by amplitude, recruitment pattern and duration across the 5 muscles (upper subscapularis, Infraspinatus, Supraspinatus, teres minor, Rhomboid) in both operated and unoperated shoulders.

SECONDARY OUTCOMES:
Tear in Rotator Cuff Muscles in both shoulders | one year post surgery
  CT Scan to evaluate rotator cuff muscles for presence or absence of any tear in operative and non-operative. If tear is present - partial or full. If full, small or (<1cm), or medium (1-3 cm_ or Large (3-5 cm) or massive (>5cm), tendon involved (supraspinatus or infraspinatus or subscapularis).
Tear in Rotator Cuff Muscles in both shoulders | two year post surgery
  CT Scan to evaluate rotator cuff muscles for presence or absence of any tear in operative and non-operative. If tear is present - partial or full. If full, small or (<1cm), or medium (1-3 cm_ or Large (3-5 cm) or massive (>5cm), tendon involved (supraspinatus or infraspinatus or subscapularis).
Fatty degeneration in Rotator Cuff Muscles in both shoulders using Goutallier Classification | one year post surgery
  CT scan to evaluate atrophy in Rotator Cuff Muscles using the Goutallier Classification System. The Classification system measures fatty tissue infiltration and has five stages, ranging from Stage 0 (normal muscle) to Stage 4 (more fat than muscle) in upper subscapularis, infraspinatus, supraspinatus, teres minor and rhomboid in both operated and unoperated shoulder.
Fatty degeneration in Rotator Cuff Muscles in both shoulders using Goutallier Classification | two year post surgery
  CT scan to evaluate atrophy in Rotator Cuff Muscles using the Goutallier Classification System. The Classification system measures fatty tissue infiltration and has five stages, ranging from Stage 0 (normal muscle) to Stage 4 (more fat than muscle) in upper subscapularis, infraspinatus, supraspinatus, teres minor and rhomboid in both operated and unoperated shoulder.
Fatty atrophy in Rotator Cuff Muscles in both shoulders | one year post surgery
  CT Scan to evaluate fatty degeneration in Rotator Cuff Muscles - present or absent in upper subscapularis, infraspinatus, supraspinatus, teres minor and rhomboid muscles in both operated and unoperated shoulders.
Fatty atrophy in Rotator Cuff Muscles in both shoulders | two year post surgery
  CT Scan to evaluate fatty degeneration in Rotator Cuff Muscles - present or absent in upper subscapularis, infraspinatus, supraspinatus, teres minor and rhomboid muscles in both operated and unoperated shoulders.

OTHER OUTCOMES:
Forward Elevation for Active Range of Motion | one year post surgery
  A physical exam will be performed on both shoulders to asses forward elevation on active range of motion using a Goniometer.
Forward Elevation for Active Range of Motion | two year post surgery
  A physical exam will be performed on both shoulders to asses forward elevation on active range of motion using a Goniometer.
Forward Elevation for Passive Range of Motion | one year post surgery
  A physical exam will be performed on both shoulders to asses forward elevation for passive range of motion using a Goniometer.
Forward Elevation for Passive Range of Motion | two year post surgery
  A physical exam will be performed on both shoulders to asses forward elevation for passive range of motion using a Goniometer.
External Rotation (side) for Passive Range of Motion | one year post surgery
  A physical exam will be performed on both shoulders to asses external rotation (side) for passive range of motion using a Goniometer.
External Rotation (side) for Passive Range of Motion | two year post surgery
  A physical exam will be performed on both shoulders to asses external rotation (side) for passive range of motion using a Goniometer.
External Rotation (side) for Active Range of Motion | one year post surgery
  A physical exam will be performed on both shoulders to asses external rotation (side) for active range of motion using a Goniometer.
External Rotation (side) for Active Range of Motion | two year post surgery
  A physical exam will be performed on both shoulders to asses external rotation (side) for active range of motion using a Goniometer.
Range of Motion in both shoulders_ Internal Rotation | one year post surgery
  Physical exam to see range of motion includes:
  Internal Rotation measured as T5 or T7 or TL or Belt or Butt or Side
Range of Motion in both shoulders_ Internal Rotation | two year post surgery
  Physical exam to see range of motion includes:
  Internal Rotation measured as T5 or T7 or TL or Belt or Butt or Side
Measurement of strength in both shoulders_Jobe's test | one year post surgery
  Measurement of Strength: measured by Isometer in Kg
Measurement of strength in both shoulders_Jobe's test | two year post surgery
  Measurement of Strength: measured by Isometer in Kg
Measurement of strength in both shoulders_External Rotation (at side) | one year post surgery
  Measurement of Strength: External Rotation (at side) measured by Isometer in Kg
Measurement of strength in both shoulders_External Rotation (at side) | two year post surgery
  Measurement of Strength: External Rotation (at side) measured by Isometer in Kg
Measurement of strength in both shoulders_Belly Press | one year post surgery
  Measurement of Strength:Belly Press measured as Positive/Negative/Unable
Measurement of strength in both shoulders_Belly Press | two year post surgery
  Measurement of Strength:Belly Press measured as Positive/Negative/Unable
Measurement of strength in both shoulders_Lift off Test | one year post surgery
  Measurement of Strength: Lift off Test as Positive/Negative/Unable
Measurement of strength in both shoulders_Lift off Test | two year post surgery
  Measurement of Strength: Lift off Test as Positive/Negative/Unable

CONTACTS AND LOCATIONS:
Overall Officials: April D Armstrong, MD, Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Penn State Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No